CLINICAL TRIAL: NCT06083519
Title: Assessment of a Novel Sound-based Treatment for Managing Distress Related to Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Lucid, Inc. (Industry); Sonova Canada Inc. (Industry); Mitacs (Industry)
Responsible Party: Principal Investigator, Brandon Paul, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: TinnitusProject_2023-333
Record Dates: First submitted 2023-09-18; First posted 2023-10-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus
Keywords: tinnitus; iso principle; artificial intelligence; auditory perception; sound therapy; neuroscience; neuromodulatory intervention; auditory beat stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- White Noise (Sham Comparator): Participants listened to white noise for 24 minutes
  Interventions: Behavioral: White Noise
- LUCID Music (Experimental): Participants listened to music chosen from the VIBE app with theta auditory beat stimulation for 24 minutes
  Interventions: Behavioral: Music and Auditory Beat Stimulation

INTERVENTIONS:
Behavioral: White Noise — This is the control condition. Listening to white noise -- participants listen to white noise for 24 minutes
  Arms: White Noise
Behavioral: Music and Auditory Beat Stimulation — Listening to music and auditory beat stimulation. The VIBE app (LUCID) incorporates theta-band (4 Hz) auditory beat stimulation and an auditory music recommendation system. Participants will listen to this music with theta auditory beat stimulation for 24 minutes.
  Other Names: LUCID Music
  Arms: LUCID Music

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of a sound-based passive treatment for reducing stress and annoyance induced by tinnitus, and how this therapy may improve tinnitus sufferers' quality of life. The main questions it aims to answer are: • [question 1: to assess the efficacy of the LUCID/VIBE in managing the tinnitus handicap (measured by the reducing of the annoyance/stress response to tinnitus) contributing to the improvement of the quality of life of people living with tinnitus] and • [question 2: assess the efficacy of LUCID/VIBE in providing temporary relief through masking, such that it results in a reduction of the perceived loudness of tinnitus]. Participants will [use the VIBE app for 24 minutes a day for a period of 4 weeks. There will be two conditions, a Noise condition (the control condition in which the investigator will administer white noise) and the VIBE condition (the treatment condition). One approach involves broad-band masking with noise (Noise Condition), while the other uses music (LUCID Condition). Implementation of the noise condition will mirror the LUCID condition in terms of ease of access, look, feel, so that one condition does not look less professional than the other. Both conditions will be administered through the same app, and only the sound conditions will differ (white noise vs. LUCID music). All participants will be exposed to both the treatment and control conditions with the order of conditions counter-balanced (i.e., a cross-over design).

DETAILED DESCRIPTION:
The current LUCID approach utilizes the VIBE app to help provide a mask for tinnitus, manage the distress related to tinnitus, and potentially dampen stress reactivity when used regularly due to the increase in parasympathetic activity. Previous findings have demonstrated that chronic tinnitus patients have elevated stress reactivity. There has also been evidence to suggest that regular music therapy interventions may enhance parasympathetic activity in the autonomic nervous system. In the past, LUCID has advanced approaches in Artificial Intelligence technology, psychology, and neuroscience to explore the potential of music to improve health and well-being. Their work to date has focused on mental health indications related to stress and anxiety. This current study differs from their previous projects because of its exploration of tinnitus rather than stress and anxiety. Their customer-facing developments have been focused on an application programming interface that has been integrated by digital-health partners and a consumer-facing app (VIBE) that has been used to support research and development. The VIBE app (LUCID) incorporates theta-band (4 Hz) auditory beat stimulation and an auditory music recommendation system. The additive effect of these elements in the treatment of acute anxiety in individuals living with moderate trait anxiety was recently demonstrated in a randomized clinical trial.

The automated music recommendation system developed by LUCID employs the iso principle along with affective classification and reinforcement learning to cultivate affect-driven personalized music sequences. The iso principal is a methodology used in music therapy to achieve mood induction that involves matching musical stimuli to a patient's current mood and gradually changing the music in the direction of their desired mood state. The iso principle has been indicated in prior research to be more effective than other musical sequences at reducing tension. The system requires that a user input their current mood using the arousal and valence dimensions of the Russell Circumplex Model. Based on this input as well as the target emotional state of calm, the machine learning algorithm within the application predicts the optimal sequence of tracks to produce mood induction in the listener from their current emotional state to the target state. This machine learning algorithm uses reinforcement learning techniques and is trained on real-world data correlating the quantitative features of musical excerpts and sequences alongside the emotional responses induced by them in listeners.

For this study. there will be two groups with 25 participants per group. For the control condition, a white-noise treatment for the noise condition will be administered. The researchers will be using an open-label randomized controlled trial study where the participants are told that the researchers are attempting to assess the effectiveness of two common interventions for tinnitus. One approach involves broad-band masking with noise (Noise Condition), while the other uses music (LUCID Condition). Implementation of the noise condition will mirror the LUCID condition in terms of ease of access, look, feel, so that one condition does not look less professional than the other. Both conditions will be administered through the same app, and only the sound conditions will differ (white noise vs. LUCID music). All participants will be exposed to both the treatment and control conditions with the order of conditions counter-balanced (i.e., a cross-over design). The LUCID treatment will be compared to the active control across 50 people. The participant is expected to engage in daily use of VIBE app at a specified time (e.g., for 24 minutes daily) and as needed to help mask symptoms of tinnitus. To minimize variability in dosage across groups, the investigators will impose daily limits and minimum adherence standards. Participants will be permitted to use the app for a maximum of 48 minutes per day (i.e., 200% of recommended dosage). Participants who use the app greater than 60 minutes (250% of recommended dosage) or less than 12 minutes per day on average (50% of recommended dosage) or who use the app on less than 75% of the trial days will be considered non-adherent and will be removed from the final sample subjected to analyses. These types of adherence boundaries are typical for decentralized clinical trials involving digital therapeutics. The VIBE app will be deployed on the participant's smartphone, and they will be instructed to use their own headphones (i.e., there is no standardization of the playback system). The app has built-in features which allow us to assess adherence to treatment. Participants in the study will experience each intervention condition for a period of 4 weeks. It is encouraged that the participants stop the study if they believe the sound therapy is exacerbating their tinnitus, their reaction to tinnitus, or negatively affecting their hearing ability.

ELIGIBILITY:
Inclusion Criteria:

* Pure-Tone Average hearing loss (500, 1000, 2000, 4000) of 30 decibels hearing loss or greater in the better ear.
* Tinnitus Handicap Index scores of 18 to 76 (mild to severe handicap).
* Self-report of chronic, non-intermittent tinnitus experienced > 3 months

Exclusion Criteria:

* Adults younger than 40 years old, or adults older than 85 years old.
* Pulsatile tinnitus (tinnitus that modulates synchronously with a participant's pulse)
* >20 dB HL difference in pure-tone average between ears
* > 80 dB HL PTA averaged across ears
* Individuals currently undergoing other tinnitus treatment programs will not be able to participate in our study. This is to ensure that our findings are accurately attributed to our App and not influenced by external factors. If someone is already receiving treatment for their tinnitus, it would be challenging to distinguish the effects of our App from their existing treatment regimen. To eliminate the possibility of such confounding factors, our team kindly asks participants to disclose if they are undergoing other treatments for tinnitus.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index | The questionnaire is administered up to two weeks pre-intervention, and again up to two weeks post-intervention measure. The measurements will be compared to see if the intervention created a change.
  The Tinnitus Functional Index is a self-report questionnaire. It is measuring the negative impact and severity of tinnitus, as well as to provide sensitive measurements to change based on treatment administration (i.e., responsiveness). This questionnaire consists of 25 questions administered in a Likert-Scale fashion ranging of a maximum value of 10 and a minimum value of 0 per question. In total, the maximum value a participant can score is 250 and the minimum is 0. A higher score (i.e., a score closer to 250), represents experiencing tinnitus at greater severity and experiencing a more negative impact from it.
36-item Short Form Health Survey | The questionnaire is administered up to two weeks pre-intervention, and again up to two weeks post-intervention measure. The measurements will be compared to see if the intervention created a change.
  The 36-item Short Form Health Survey is a measurement tool used to assess subjective quality of life. A study has found this tool to be reliable and valid.

SECONDARY OUTCOMES:
Visual Analogue System | Up to 48 hours after each usage.
  Our visual analogue scale measures tinnitus annoyance using a continuous slider scale on a computer or touch-screen interface. The bottom of the scale (to the left) is "Not annoying" and the top of the scale (to the right) is "Highest possible annoyance".

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Paul, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators are going to register the project on Open Science Framework and will make all elements of individual participant data open to the public post-data collection and after de-identification.
Supporting Information: Study Protocol, ICF
Time Frame: Data are available now and will be for 7 years post-data collection completion.
Access Criteria: There are no specific access criteria for the individual participant data on the Open Science Framework. It is freely and openly available to anyone.

REFERENCES:
- [Background] Aazh H, Salvi R. The Relationship between Severity of Hearing Loss and Subjective Tinnitus Loudness among Patients Seen in a Specialist Tinnitus and Hyperacusis Therapy Clinic in UK. J Am Acad Audiol. 2019 Sep;30(8):712-719. doi: 10.3766/jaaa.17144. Epub 2018 Nov 8. PMID 30403955
- [Background] Garcia-Argibay M, Santed MA, Reales JM. Efficacy of binaural auditory beats in cognition, anxiety, and pain perception: a meta-analysis. Psychol Res. 2019 Mar;83(2):357-372. doi: 10.1007/s00426-018-1066-8. Epub 2018 Aug 2. PMID 30073406
- [Background] Gopinath B, McMahon CM, Rochtchina E, Karpa MJ, Mitchell P. Risk factors and impacts of incident tinnitus in older adults. Ann Epidemiol. 2010 Feb;20(2):129-35. doi: 10.1016/j.annepidem.2009.09.002. PMID 20123163
- [Background] Hall DA, Haider H, Szczepek AJ, Lau P, Rabau S, Jones-Diette J, Londero A, Edvall NK, Cederroth CR, Mielczarek M, Fuller T, Batuecas-Caletrio A, Brueggemen P, Thompson DM, Norena A, Cima RF, Mehta RL, Mazurek B. Systematic review of outcome domains and instruments used in clinical trials of tinnitus treatments in adults. Trials. 2016 Jun 1;17(1):270. doi: 10.1186/s13063-016-1399-9. PMID 27250987
- [Background] Hullfish J, Sedley W, Vanneste S. Prediction and perception: Insights for (and from) tinnitus. Neurosci Biobehav Rev. 2019 Jul;102:1-12. doi: 10.1016/j.neubiorev.2019.04.008. Epub 2019 Apr 15. PMID 30998951
- [Background] Mallik A, Russo FA. The effects of music & auditory beat stimulation on anxiety: A randomized clinical trial. PLoS One. 2022 Mar 9;17(3):e0259312. doi: 10.1371/journal.pone.0259312. eCollection 2022. PMID 35263341
- [Background] McConnell PA, Froeliger B, Garland EL, Ives JC, Sforzo GA. Auditory driving of the autonomic nervous system: Listening to theta-frequency binaural beats post-exercise increases parasympathetic activation and sympathetic withdrawal. Front Psychol. 2014 Nov 14;5:1248. doi: 10.3389/fpsyg.2014.01248. eCollection 2014. PMID 25452734
- [Background] Nondahl DM, Cruickshanks KJ, Dalton DS, Klein BE, Klein R, Schubert CR, Tweed TS, Wiley TL. The impact of tinnitus on quality of life in older adults. J Am Acad Audiol. 2007 Mar;18(3):257-66. doi: 10.3766/jaaa.18.3.7. PMID 17479618
- [Background] Zhang Y, Qu B, Lun SS, Guo Y, Liu J. The 36-item short form health survey: reliability and validity in Chinese medical students. Int J Med Sci. 2012;9(7):521-6. doi: 10.7150/ijms.4503. Epub 2012 Aug 27. PMID 22991490
- [Background] Rider, M. S. (1985). Entrainment mechanisms are involved in pain reduction, muscle relaxation, and musicmediated imagery. Journal of Music Therapy, 22(4), 183-92. doi: 10.1093/jmt/22.4.183.
- [Background] Heiderscheit, A., Madson, A. (2015). Use of the iso principle as a central method in mood management: A music psychotherapy clinical case study. Music Therapy Perspectives, 33(1), 45-52.
- [Background] Labbé A, McMahon, Z., & Thomson, Z. (2021). Music as Medicine: LUCID Science + Technology White Paper. [White Paper]. Available online at https://uploads ssl.webflow.com/60b8a3f8bd91d547f8a453dc/614e1cead49a3cadb1880924_Whitepaper%20- %20Public-Facing.pdf
- [Background] Remmington NA, Fabrigar LR, Visser PS. Reexamining the circumplex model of affect. J Pers Soc Psychol. 2000 Aug;79(2):286-300. doi: 10.1037//0022-3514.79.2.286. PMID 10948981
- [Background] Sindhusake D, Golding M, Newall P, Rubin G, Jakobsen K, Mitchell P. Risk factors for tinnitus in a population of older adults: the blue mountains hearing study. Ear Hear. 2003 Dec;24(6):501-7. doi: 10.1097/01.AUD.0000100204.08771.3D. PMID 14663349
- [Background] Starcke K, Mayr J, von Georgi R. Emotion Modulation through Music after Sadness Induction-The Iso Principle in a Controlled Experimental Study. Int J Environ Res Public Health. 2021 Nov 26;18(23):12486. doi: 10.3390/ijerph182312486. PMID 34886210
- [Background] Vernon D, Peryer G, Louch J, Shaw M. Tracking EEG changes in response to alpha and beta binaural beats. Int J Psychophysiol. 2014 Jul;93(1):134-9. doi: 10.1016/j.ijpsycho.2012.10.008. Epub 2012 Oct 17. PMID 23085086